CLINICAL TRIAL: NCT07074639
Title: S.M.A.R.T: A Pragmatic Randomised Controlled Trial of Personalized Cognitive-Motor Exergame Training in Frail Community-Dwelling Adults
Brief Title: Cognitive-Motor Exergame Training in Frail Adults
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eleftheria Giannouli (Other)
Responsible Party: Sponsor-Investigator, Eleftheria Giannouli, Principal Investigator, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S.M.A.R.T.
Record Dates: First submitted 2025-06-15; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Aging; Frailty
Keywords: Frailty; Aging; Cognitive training; Physical activity; Home-based intervention; exergames; dual-task training; fall-prevention
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a single-blind (assessor blind) international, pragmatic, two-arm randomized controlled trial (RCT) conducted in five countries/trial sites: ETH Zurich/University Hospital Zurich (Zurich, Switzerland), Don Carlo Gnocchi Foundation (Milan, Italy), Alma Mater Europaea University/General Hospital Izola (Koper/Izola, Slovenia), Materia Agecare (Nicosia, Cyprus), and Saint Vincent De Paul long term care facility (Luqa, Malta). The study has an intervention group (IG) and a control group (CG) and will consist of 12 weeks of intervention with 12 weeks of follow-up period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the IG will receive personalized cognitive-motor training in their home environment. The simultaneous cognitive-motor training in this study will be delivered using the exergame platform "Senso Flex" by Dividat (Dividat AG, Schindellegi, Switzerland). The first session will be supervised by an investigator. Afterwards, participants will continue the training independently at home, with remote supervision and guidance. Participants will be recommended to train 5 times per week for 30 minutes in each session over a 12-week period. Weekly game play will be 150 min to help ensure equal doses of training between IG and CG. The training plan for each participant will be tailored to ensure a progressive and personalized approach. Besides, participants of the intervention group will participate in 3 assessment sessions: (1) T1 (baseline assessments), (2) T2 (post-intervention, after training period), (3) T3 (follow-up assessment).
  Interventions: Other: Personalized, home-based motor-cognitive exergame training
- Control Group (Active Comparator): Participants in the CG will receive the evidence-based OEP on fall prevention. Like for the IG, participants of the CG will be recommended to train 5 times per week for 30 minutes in each session. The training will be conducted over a 12-week period, with a total weekly duration of 150 minutes. The first session will be supervised by an investigator. The program will be implemented in the form of a booklet, designed to provide a comprehensive guide for improving balance, strength, and overall physical function. Like the IG, the participants of the control group will also participate in 3 assessment sessions: (1) T1 (baseline assessments), (2) T2 (post-intervention, after training period), (3) T3 (follow-up assessment).
  Interventions: Other: Otago Exercise Program

INTERVENTIONS:
Other: Personalized, home-based motor-cognitive exergame training — The simultaneous cognitive-motor training in this study will be delivered using the exergame platform "Senso Flex" by Dividat (Dividat AG, Schindellegi, Switzerland), which is a pressure-sensitive foldable mat that connects to standard televisions (or any big screen). Games will be allocated across three primary domains: cognition (consisting of five sub-domains), balance (consisting of four sub-domains) and endurance. The five sub-domains of cognition are visuospatial orientation (Cognition A), memory (Cognition B), response inhibition (Cognition C), choice reaction time (Cognition D) and task switching (Cognition E). The four sub-domains of balance are mediolateral weight-shifting (Balance A), multidimensional weight-shifting (Balance B), free walking/stepping (Balance C) and mediolateral stepping (Balance D). The training sessions will be personalized in terms of difficulty level.
  Arms: Intervention Group
Other: Otago Exercise Program — Participants in the CG will receive the evidence-based OEP on fall prevention. The OEP was selected as an active control to mirror usual care in real-world clinical settings and support the pragmatic nature of our study design. The program will be implemented in the form of a booklet, designed to provide a comprehensive guide for improving balance, strength, and overall physical function. Specifically tailored for older adults, the program includes a variety of exercises targeting key areas such as lower limb strength, balance, and flexibility. It features step-by-step instructions, illustrations, and tips to ensure exercises are performed safely and effectively.
  Arms: Control Group

SUMMARY:
This international multicentre pragmatic randomized controlled trial (RCT) aims to evaluate the effectiveness of personalized, home-based cognitive-motor training using exergames in improving cognitive and motor functions in frail adults. A total of 344 frail participants from five European countries will be enrolled. Participants in the intervention group will engage in a personalized exergame program, while the control group will follow the Otago Exercise Program. Both groups will undergo 12 weeks of training. The primary outcome is balance, a critical component of functional independence and fall prevention, and a common denominator affected in both physical and cognitive frailty. Secondary outcomes including cognitive and motor fall-risk factors, fall incidence, cost-effectiveness, and psychosocial outcomes.

DETAILED DESCRIPTION:
The global population is aging rapidly, with those aged 60+ expected to double by 2050. While longevity is increasing due to better healthcare and living conditions, this shift poses major challenges, frailty being a key concern. Affecting 5%-58% of older adults, frailty compromises independence, quality of life, and healthcare systems. It is a dynamic condition marked by vulnerability to stressors and can appear as physical, cognitive, or combined frailty.

Physical frailty is well-studied, often defined by low gait speed, fatigue, weakness, weight loss, and reduced activity, but broader health indicators are also used. Cognitive frailty, recognized more recently, is defined as the co-existence of physical frailty and cognitive impairment without dementia. It may signal early dementia risk and greater susceptibility to adverse outcomes.

A core feature of frailty is balance dysfunction, caused by impairments in sensory, cognitive, and motor systems. This is especially problematic during dual tasks, like walking while talking, where attention is divided. Such deficits increase fall risk and accelerate cognitive and physical decline.

Traditional fall prevention emphasizes strength and balance, often overlooking cognitive factors. Yet, evidence shows that motor and cognitive systems are linked, and dual-task training can enhance both domains. Cognitive-motor training, which integrates cognitively demanding tasks into physical exercises, offers a promising dual-domain intervention by leveraging shared brain networks and promoting neuroplasticity.

While effective, most cognitive-motor programs are delivered in person and rarely tailored to individual frailty profiles. Personalized, home-based programs could offer better results through tailored challenge and engagement. Exergames, interactive digital games with physical and cognitive components, show promise as customizable, engaging tools for such training. However, few have integrated both domains simultaneously in frail adults.

This study aims to assess a 12-week, home-based personalized cognitive-motor training program against the Otago Exercise Program (OEP) in frail older adults. Outcomes include physical and cognitive fall-risk factors, fall incidence, quality of life, and physical activity. The hypothesis is that the personalized cognitive-motor program will lead to greater improvements and may offer an effective, scalable solution to reduce falls and promote independence in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and older
* Fried Frailty Phenotype score 3 or higher and/or MoCA score between 10-25
* Must be able to give informed consent
* Access to internet and a TV/large screen at home

Exclusion Criteria:

* Mobility limitations (e.g., severe arthritis or lower extremity amputation)
* Cognitive limitations (e.g., advanced Alzheimer's disease, frontotemporal/Lewy body/vascular dementia)
* Sensory limitations (e.g., color-blindness, complete hearing loss and neuropathy causing significant loss of sensation)
* Psychiatric limitations (e.g., acute, or uncontrolled affective disorders)
* Comorbidities that would impair their ability to engage in the training
* Simultaneous participation in other clinical trials/intervention studies
* Inability to understand game instructions and play the games safely, based on judgement of a therapist

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Balance | The primary outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The primary outcome measure is balance, which will be assessed by using Berg Balance Scale (BBS). Balance is the ability to maintain stability and control of the body during everyday activities or movements, encompassing both static and dynamic balance. By focusing on balance, the aim is to gain insights into frail adults' ability to remain autonomous and prevent or slow down further frailty-related decline. The BBS has been selected for its proven reliability and validity in assessing balance and predicting fall risk in this population. BBS is a quantitative tool used to assess a patient's ability, or inability, to maintain balance safely during a series of predetermined activities. The scale consists of 14 items, each rated on a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of functional ability and 4 representing the highest.

SECONDARY OUTCOMES:
Dynamic balance | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The Four-Square Step Test (FSST) will be used to measure dynamic balance by timing (in seconds) how long a subject takes to step forward, backward, and sideways through four floor-marked squares in a specific sequence and then reverse back to the starting position.
Lower extremity function | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  Lower extremity function will be evaluated using the Short Physical Performance Battery (SPPB). The SPPB includes three timed tasks: maintaining static balance in three-foot positions, walking 4 meters to assess gait speed, and performing five consecutive sit-to-stand movements. Minimum score: 0, Maximum score: 12.
  Higher scores indicating better lower extremity function.
Functional Mobility and Balance in Single Task | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  Functional mobility and balance will be evaluated in single task using the Timed Up and Go (TUG) test. The TUG test measures the time needed to stand up, walk 3 meters at a normal pace, turn, return to the chair, and sit down (in seconds).
Functional Mobility and Balance in Dual-Task | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  Functional mobility and balance in dual-task will be evaluated using the Timed Up and Go (TUG) test in dual task (DT) conditions - here a cognitive task, in which participants will be instructed to count backwards from 100, subtracting 2 successively, will be added to the main TUG task. Outcome of this test is duration. Higher values indicate lower performance.
Dual-Task Costs | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  Dual-task cost (DTC) will be calculated using the values of the TUG test in single task and the TUG test in dual-task using the formula:
  DTC (%) = [(Single-task performance - Dual-task performance) / Single-task performance] * 10
Functional capacity | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The 6-Minute Walk Test (6MWT) will measure functional capacity by recording the distance walked (in meters) at a brisk, self-paced speed over six minutes, reflecting the integrated physiological response of multiple systems.
Performance Fatigability | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  Performance fatigability, which objectively captures how physical performance worsens over time, offering insights into endurance and fall risk, is then calculated as the ratio (%) of mean walking speed over six minutes (V6 min) to the mean speed of the first two minutes (V2 min), divided by the total distance (meter) and scaled by 1000 .
Response inhibition (reaction time) | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The go/no-go test measures response inhibition by evaluating (amongst other measures) reaction time (in milliseconds) as participants respond to "go" stimuli and suppress responses to "no-go" stimuli. All cognitive assessments will be conducted using PsyToolkit, an open-source platform widely used for implementing computerized cognitive tasks in research settings.
Response inhibition (error rate) | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The go/no-go test measures response inhibition by evaluating (amongst other measures) errors as participants respond to "go" stimuli and suppress responses to "no-go" stimuli. All cognitive assessments will be conducted using PsyToolkit, an open-source platform widely used for implementing computerized cognitive tasks in research settings.
Cognitive flexibility (reaction time) | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The multitasking test evaluates cognitive flexibility by requiring participants to switch between shape and filling tasks based on stimulus location, measuring (amongst other measures) reaction time (in milliseconds). All cognitive assessments will be conducted using PsyToolkit, an open-source platform widely used for implementing computerized cognitive tasks in research settings.
Cognitive flexibility (error rate) | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The multitasking test evaluates cognitive flexibility by requiring participants to switch between shape and filling tasks based on stimulus location, measuring (amongst other measures) errors. All cognitive assessments will be conducted using PsyToolkit, an open-source platform widely used for implementing computerized cognitive tasks in research settings.
Psychomotor Speed | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The Deary-Liewald Task assesses (amongst other measures) reaction times (in milliseconds) by measuring participants' responses to stimuli in a simple reaction time task or their ability to select the correct key in a choice reaction time task. All cognitive assessments will be conducted using PsyToolkit, an open-source platform widely used for implementing computerized cognitive tasks in research settings.
Psychomotor errors | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The Deary-Liewald Task assesses (amongst other measures) errors by measuring participants' responses to stimuli in a simple reaction time task or their ability to select the correct key in a choice reaction time task. All cognitive assessments will be conducted using PsyToolkit, an open-source platform widely used for implementing computerized cognitive tasks in research settings.
Sustained attention and response inhibition (reaction time) | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The sustained attention to response task measures sustained attention and response inhibition by requiring responses to digits from '1' to '9' except for '3', assessing (amongst other measures) reaction time (in milliseconds). All cognitive assessments will be conducted using PsyToolkit, an open-source platform widely used for implementing computerized cognitive tasks in research settings.
Sustained attention and response inhibition (error rate) | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The sustained attention to response task measures sustained attention and response inhibition by requiring responses to digits from '1' to '9' except for '3', assessing (amongst other measures) errors. All cognitive assessments will be conducted using PsyToolkit, an open-source platform widely used for implementing computerized cognitive tasks in research settings.
Fall incidence | Fall history will be collected at most 1 week prior to starting the intervention. Fall incidence will be collected continuously throughout the intervention, as well as during the 12 weeks post-intervention.
  Falls will be monitored through detailed records of falls within the past 12 months. Monitoring will involve tracking of fall frequency through regular telephone calls during which participants will be asked to report the number of falls they have experienced since the last contact (conducted weekly for the first three weeks and biweekly thereafter).
Fear of falling | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  The Falls Efficacy Scale - International will be used to assess participants' confidence in their ability to avoid falls during different activities. The scale goes from 16 points (minimum value, no fear of falling) to 64 points (maximum value, severe concern about falling).
Quality of life parameters | This outcome will be measured at most 1 week prior to starting the intervention, one week after finishing the intervention and then again 12 weeks after the end of the intervention.
  Quality of life will be measured using the EuroQol 5-Dimension 5-Level Questionnaire, which evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Participants will be asked to report the level of difficulties they encounter in these dimensions, choosing from 5 levels (1 being no problems encountered, 5 being extreme problems in this dimension).
  Furthermore the EuroQol VAS (visual analog scale) will be used. Participants will rate their health-related quality of life on a scale from 0-100, with the lowest value meaning the worst health state they can imagine, and the highest value meaning the best health state they can imagine.
Exergame Enjoyment Questionnaire | This outcome will be measured at most 1 week after the end of the intervention.
  The exergame enjoyment questionnaire assesses enjoyment of the exergame intervention at the intervention group (IG). The minimum score is 20 points and the maximum score is 100 points. Higher scores are better, indicating more enjoyment.
Usability | This outcome will be measured at most 1 week after the end of the intervention.
  The System Usability Scale (SUS) will be used to assess usability of the cognitive-motor exergame training system within IG. Higher scores indicate higher usability. The minimum score is 0 points and the maximum score is 100 points. A higher score is better and indicates better usability.
Adherence | This outcome will be recorded continuously throughout the intervention period, namely in the weeks 1, 2 , 3, 5, 7, 9, 11, and 12 of the intervention.
  Adherence will be assessed based on the weekly training duration, measured as the total time spent on training each week (in minutes). This data will be recorded and displayed in the rehabilitation cockpit (Dividat Manager system). The adherence rate will be calculated as the number and duration of completed training sessions relative to the recommended number and duration, expressed as a percentage (%). The regular telephone calls will also be used to enhance adherence to the training program. Adherence in the CG will be monitored through regular phone calls, as in the IG, and paper-based training logs, which participants will return at post-intervention assessment visit.
Level of assistance | This outcome will be measured at most 1 week before the intervention starts, then continuously throughout the intervention period and again 12 weeks after the end of the intervention.
  The level of assistance required by the participant, measured in weekly hours of formal or informal caregiving, as well as information related to physical and cognitive activities and interventions will be collected through an ad hoc questionnaire during regular telephone calls, to provide the data needed to perform the cost-effectiveness analysis. The lowest level is "no assistance" and the highest level is "full assistance".
Adverse events | This outcome will be measured starting from at most 1 week before the intervention, throughout the intervention until the final measurement 12 weeks after the end of the intervention.
  Total number of (Serious) Adverse Events (SAE/AE).
Attrition rate | This outcome will be measured starting from at most 1 week before the intervention, throughout the intervention until the final measurement 12 weeks after the end of the intervention.
  Number of drop-outs of patients included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eleftheria Giannouli, PhD, Principal Investigator — ETH Zurich
Locations (1):
- Institute of Human Movement Sciences and Sport, ETH Zürich, Zurich, Switzerland

REFERENCES:
- [Background] Seinsche J, Kyprianou E, de Bruin ED, Saibene E, Rizzo F, Carpinella I, Lutz L, Ferrarin M, Villa R, Chrysostomou S, Moza S, Giannouli E. Discriminative ability of instrumented cognitive-motor assessments to distinguish fallers from non-fallers. Geroscience. 2025 Feb;47(1):1139-1150. doi: 10.1007/s11357-024-01313-x. Epub 2024 Aug 9. PMID 39120688
- [Background] Seinsche J, de Bruin ED, Saibene E, Rizzo F, Carpinella I, Ferrarin M, Ifanger S, Moza S, Giannouli E. Feasibility and Effectiveness of a Personalized Home-Based Motor-Cognitive Training Program in Community-Dwelling Older Adults: Protocol for a Pragmatic Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 9;12:e49377. doi: 10.2196/49377. PMID 37943591
- [Background] Rainero I, Summers MJ, Monter M, Bazzani M, Giannouli E, Aumayr G, Burin D, Provero P, Vercelli AE; My-AHA Consortium. The My Active and Healthy Aging ICT platform prevents quality of life decline in older adults: a randomised controlled study. Age Ageing. 2021 Jun 28;50(4):1261-1267. doi: 10.1093/ageing/afaa290. PMID 33480986
- [Background] Glatt RM, Patis C, Miller KJ, Merrill DA, Stubbs B, Adcock M, Giannouli E, Siddarth P. The "FitBrain" program: implementing exergaming & dual-task exercise programs in outpatient clinical settings. Front Sports Act Living. 2024 Dec 6;6:1449699. doi: 10.3389/fspor.2024.1449699. eCollection 2024. PMID 39712081
- [Background] Seinsche J, de Bruin ED, Saibene E, Rizzo F, Carpinella I, Ferrarin M, Moza S, Ritter T, Giannouli E. A Newly Developed Exergame-Based Telerehabilitation System for Older Adults: Usability and Technology Acceptance Study. JMIR Hum Factors. 2023 Dec 7;10:e48845. doi: 10.2196/48845. PMID 38060283
- [Background] Seinsche J, de Bruin ED, Carpinella I, Ferrarin M, Moza S, Rizzo F, Salatino C, Giannouli E. Older adults' needs and requirements for a comprehensive exergame-based telerehabilitation system: A focus group study. Front Public Health. 2023 Jan 11;10:1076149. doi: 10.3389/fpubh.2022.1076149. eCollection 2022. PMID 36711352
- [Background] Bernardes RA, Giannouli E, Neves H, Parola V. Editorial: User-centered technology for exercise optimization in older adults. Front Sports Act Living. 2025 Feb 4;7:1558979. doi: 10.3389/fspor.2025.1558979. eCollection 2025. No abstract available. PMID 39968188
- [Background] Buttiker J, Marks D, Hanke M, Ludyga S, Marsico P, Eggimann B, Giannouli E. Cognitive-motor exergame training on a labile surface in stroke inpatients: study protocol for a randomized controlled trial. Front Neurol. 2024 Jun 19;15:1402145. doi: 10.3389/fneur.2024.1402145. eCollection 2024. PMID 38966081
- [Background] Jaggi S, Wachter A, Adcock M, de Bruin ED, Moller JC, Marks D, Schweinfurther R, Giannouli E. Feasibility and effects of cognitive-motor exergames on fall risk factors in typical and atypical Parkinson's inpatients: a randomized controlled pilot study. Eur J Med Res. 2023 Jan 16;28(1):30. doi: 10.1186/s40001-022-00963-x. PMID 36647177
- [Background] Altorfer P, Adcock M, de Bruin ED, Graf F, Giannouli E. Feasibility of Cognitive-Motor Exergames in Geriatric Inpatient Rehabilitation: A Pilot Randomized Controlled Study. Front Aging Neurosci. 2021 Nov 29;13:739948. doi: 10.3389/fnagi.2021.739948. eCollection 2021. PMID 34912206